CLINICAL TRIAL: NCT06000839
Title: A Prospective, Open Study on the Safety and Effectiveness of CELLBOOSTER® Lift (Stabilized Booster Complex Using CHAC Technology) on Healthy Subjects
Brief Title: A Safety and Effectiveness Study of CELLBOOSTER® Lift (Stabilized Booster Complex Using CHAC Technology)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suisselle (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21E4451
Record Dates: First submitted 2023-05-08; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Skin Fold; Skin Laxity; Skin Texture Disorder; Skin Depression; Skin Dryness; Hyperpigmentation; Atrophic Scar; Striae Distensae; Oxidative Stress
Keywords: Skin Fold; Skin Laxity; Skin Depression; Skin Texture Disorder; Skin Dehydration; Skin Dryness; Skin Quality; Microvascular Circulation; Hyperpigmentation; Oxidative Stress; Atrophic Scar; Striae Distensae; Acne Scars - Mixed Atrophic and Hypertrophic; Epidermis; Dermis; Aesthetic Effect; Aesthetic; Face Treatment; Injection; Micro Papula; Papula; Injection Protocol; Healthy Subjects; Adverse Events; Adverse Effects; Efficacy; Safety; Performance; CELLBOOSTER; Lift; SUISSELLE
MeSH Terms: conditions — Cutis Laxa; Hyperpigmentation; Striae Distensae; Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CELLBOOSTER® Lift (Experimental)
  Interventions: Device: (D0) Intradermal injection - micropapula technique; Device: (D14) Intradermal injection - micropapula technique; Device: (D28) Intradermal injection - micropapula technique

INTERVENTIONS:
Device: (D0) Intradermal injection - micropapula technique — First injection of the product (3ml) in the medium and lower third of the face (whole face excepted forehead)
Device: (D14) Intradermal injection - micropapula technique — Second injection of the product (3ml) in the medium and lower third of the face (whole face excepted forehead)
Device: (D28) Intradermal injection - micropapula technique — Third injection of the product (3ml) in the medium and lower third of the face (whole face excepted forehead)

SUMMARY:
The current post-market clinical investigation has been designed to evaluate the efficacy and safety of CELLBOOSTER® Lift, a HA-based product marketed by SUISSELLE SA. For this purpose, healthy subjects with signs of skin aging with mild to moderate wrinkles, skin laxity, dry and dull skin on the face, received a 3-session treatment and were followed-up over a 4-month period after the initial injection.

Several objective measurements of skin quality were performed with different parameters: skin elasticity, density, dryness, microcirculation, wrinkles, color/homogeneity. Clinical improvement was also evaluated, as well as subject and investigator satisfactions.

The safety of the injections was also followed with injection site reactions and adverse events collection.

DETAILED DESCRIPTION:
With age and UV exposure, skin undergoes morphologic and mechanical changes that manifest as wrinkling, sagging, loss of elasticity and dryness. In particular, decreased synthesis of collagen and elastin and their increased degradation reduced proliferative capacity of fibroblasts. Moreover, the perturbations in the organisation of elastic fibre network lead to alterations in the mechanical properties of the skin with reduced resilience and elasticity. Advances in the knowledge of the biochemical mechanisms associated with ageing have led to the development of different approaches to reduce and repair its untoward effects, particularly by using minimally invasive procedures. Originally developed to treat vascular and lymphatic disorders, mesotherapy has recently been used for skin rejuvenation.

Mesotherapy consists of the stimulation of skin biorejuvenation via minimally invasive epidermis or intradermal injections of biologically active substances. The injected ingredients are released over a prolonged period of time into the surrounding tissues, with a depot-like effect. Among the products available for skin rejuvenation by mesotherapy, hyaluronic acid (HA) plays an important role in the moisturization due to its high ability to attract water molecules. Given all the above, HA was a clear natural candidate for such applications, and non-crosslinked HA gels are by far the most popular compounds employed for mesotherapy, both alone and in combination with other molecules. Mesotherapy with HA aids in restoring cutaneous metabolic function, water retention and elasticity, with an altogether improvement in the visible signs of photoaging. The efficacy of non-crosslinked HA injections for the treatment of photoaged skin has been widely reported.

HA-based injections may be supplemented with other active ingredients for additional, synergistic benefits, on condition the compounds be biocompatible and absorbable, such as vitamins, antioxidants and/or amino acids.

Clinical experience of skin rejuvenation by HA-based mesotherapy suggests this technique is safe inasmuch as it is performed by a trained physician, who follows safe-injection practices with appropriate aseptic techniques to prevent, among other, the risk of infection related to inadequate safety measures. Furthermore, several studies suggest mesotherapy can improve skin hydration, firmness and viscoelastic properties. Usually, this type of treatment includes an intensive course with 3 treatments with 2-3 weeks interval, followed by a support course with one treatment per month. The number of treatments needed will depend on the patients (age, skin condition, answer to initial treatment,….).

SUISSELLE has marketed in 2021 the HA-based product CELLBOOSTER® Lift (CBL). CBL consists in a stabilized HA complex with amino acids and vitamins for injection in the epidermis or dermis.

The current post-market clinical investigation is designed to evaluate the efficacy and safety of CBL. For this purpose, healthy subjects with signs of skin aging with mild to moderate wrinkles, skin laxity, dry and dull skin on the face, received a 3-session treatment and were followed-up over a 4-month period after the initial injection.

Several objective measurements of skin quality were performed with different parameters: skin elasticity, density, dryness, microcirculation, wrinkles, color/homogeneity. Clinical improvement was also evaluated, as well as subject and investigator satisfactions.

The safety of the injections was also followed with injection site reactions and adverse events collection.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Phototype II to III
* Subject with signs of cutaneous ageing on the face with mild to moderate wrinkles, skin laxity, dry and dull skin on face.
* Subject with a skin hydration rate on cheekbones < 60 UA, measured with Corneometer®.
* Subject looking for an improvement using an aesthetic procedure.
* Subject willing to abstain from other facial aesthetic procedure in the full face through the entire study duration.
* Subject having given their free, express, and informed consent.
* Subject psychologically able to understand the information related to the study, and to give their written informed consent.
* Subject registered with a social security scheme.
* Female of childbearing potential must use a medically accepted contraceptive method since at least 12 weeks before the beginning of the study and throughout the study.
* Female subjects of childbearing potential must have a negative pregnancy test at the inclusion.

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study.
* Woman menopaused from less than 1 year or in perimenopause, without hormonal treatment.
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship.
* Subject in a social or sanitary establishment.
* Subject participating to another research on human beings or being in an exclusion period for a previous study.
* Subject having received a total of 4.500 euros as compensations for their participation in research involving human beings in the last 12 months, including their participation in the present study.
* Intensive exposure to sunlight or UV-rays within the previous month and/or planning to do so during the study.
* Subject with a tattoo, a scar, moles or too many hairs or anything on the face which may interfere with the study at the investigator appreciation.
* Subject having resorbable filling product (e.g., hyaluronic acid) injections, a laser treatment, an ultrasound-based treatment, a dermabrasion, a deep chemical peeling or other ablative procedure on the face within the past 12 months prior to study start and a facial surgery in the past 2 years
* Subjects having received botulinum toxin in the face within the 9 previous months.
* Subject having received mesotherapy products in the face within the 3 previous months.
* Subject having done a superficial or medium peeling or a superficial scrub on the face within the 2 previous months.
* Subject using cosmetic products with alpha hydroxy acids (AHA).
* Subject with subcutaneous retaining structure on the face (meshing, threads, gold strand).
* Subject having received injections of permanent (e.g., acrylate polymers, silicone, polytetrafluoroethylene) or semi-permanent filling on the face (L Polylactic acid, Calcium Hydroxyapatite...).
* Subject with an excessive consumption of alcohol (more than 2 glasses of wine per day) and/or tobacco (more than 10 cigarettes per day).
* Subject with unstable weight or planning to do a dietary regime during the study.
* Subject with a BMI>30.
* Subject with ongoing and/or uncontrolled and/or recently recovered (<6 months) depression or psychiatric disorders or any other disorder that may pose a health risk to the subject in the study and/or may have an impact on the study assessments.
* Subject with severe, ongoing and uncontrolled diseases such as malignancy or history of malignancy, type I diabetes, liver failure, renal failure, lung/heart disease, neoplasia, malignant blood disease, tumor, HIV, or other major disease (e.g., systemic fungal infection).
* Subject with recurrent porphyria, coronary insufficiency, ventricular rhythm disorders, severe hypertension, obstructive cardiomyopathy, hyperthyroidism.
* Subject with any skin or systemic disease (acute and/or chronic), in the previous year, likely to interfere with the measured parameters or to put the subject to an undue risk.
* Subject with known history of or suffering from autoimmune disease and/or immune deficiency.
* Subject with current cutaneous inflammatory or infectious processes (e.g., acne, herpes, mycosis, papilloma, chronic eczema, atopic dermatitis …), abscess, unhealed wound, or a cancerous or precancerous lesion on the face.
* Subject with multiple allergies, anaphylactic shock history, evolutive allergic pathologies.
* Subject having history of allergy or hypersensitivity to one of the components of the tested device
* Subject having history of hypersensitivity to the antiseptic solution, to lidocaine and/or prilocaine or local anesthetics of amide type or one of the excipients of EMLA 5% cream.
* Subject predisposed to keloids or hypertrophic scarring.
* Subject with coagulation and/or homeostasis disorders.
* Subject with pigmentation disorders (vitiligo, melasma,….).
* Subject under anti-coagulant treatment (such as aspirin, nonsteroidal anti-inflammatory drugs) or treatment liable to interfere with the healing process or hemostasis, during the previous month and during the study.
* Subject receiving any treatment that, in the opinion of the clinical investigator, may interfere with test results or put the subject to undue risk.
* Subject undergoing a topical (on the face) or systemic treatment:

  * anti-inflammatory medication during the previous 2 weeks and during the study;
  * anti-histaminics during the previous 3 days;
  * immunosuppressors and/or corticoids during the 4 previous weeks and during the study;
  * retinoids during the 6 previous months and during the study.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of epidermis hydration higher than 2 AU | Baseline, Day 42
  Measured with a Corneometer®

SECONDARY OUTCOMES:
Change from baseline of epidermis hydration | Baseline, Day 84
  Measured with a Corneometer®
Change from baseline of cutaneous firmness | Baseline, Day 42 and Day 84
  Based on the skin deformation curve obtained with a Cutometer®, the cutaneous firmness, or final deformation (Uf, in mm), is the maximal amplitude of the deformation
Change from baseline of the elasticity | Baseline, Day 42 and Day 84
  Based on the skin deformation curve obtained with a Cutometer®, the elasticity is the ratio between various elongation amplitudes (Ur/Ue, Uv/Ue, Ua/Uf)
Change from baseline of the tonicity | Baseline, Day 42 and Day 84
  Based on the skin deformation curve obtained with a Cutometer®, the tonicity, or elastic return (Ur, in mm) is the immediate retractation of the skin after the suction
Change from baseline of the suppleness | Baseline, Day 42 and Day 84
  Based on the skin deformation curve obtained with a Cutometer®, the suppleness (Ue, in mm) is the immediate elongation of the skin during the suction
Change from baseline of skin density | Baseline, Day 42 and Day 84
  Measured with Dermascan®
Change from baseline of skin microcirculation | Baseline, Day 42 and Day 84
  Measured with Laser Doppler
Change from baseline of skin wrinkles parameters | Baseline, Day 42 and Day 84
  Measured with a fringe projection system
Change from baseline of skin color parameters | Baseline, Day 42 and Day 84
  Measured on 2D photographies
Percentage of subjects with a GAIS score "improved", "much improved", or "very much improved" (investigator) | Baseline, Day 42 and Day 84
  The Global Aesthetic Improvement Scale (GAIS) is a five-point scale for assessing global aesthetic improvement in appearance compared to pretreatment. This change has been assessed by the investigator.
Percentage of subjects with a GAIS score "improved", "much improved", or "very much improved" (subjects) | Baseline, Day 42 and Day 84
  The Global Aesthetic Improvement Scale (GAIS) is a five-point scale for assessing global aesthetic improvement in appearance compared to pretreatment. This change has been assessed by the subjects.
Degree of satisfaction of the subjects | Baseline, Day 42 and Day 84
  Satisfaction assessed through the answers to a subjective evaluation questionnaire.
Degree of satisfaction of the injectors | After each injection (Day 0, Day 14 and Day 28)
  Satisfaction assessed through the answers to a subjective evaluation questionnaire completed for each subjects after injection. Satisfaction assessed on a scale from "Very dissatisfied" to "Very satisfied".

OTHER OUTCOMES:
Collection of reactions at injection sites and adverse events (safety endpoint) | Baseline, Day 0, Day 14, Day 28, Day 42, Day 84
  Evaluation of the injection site reactions by the injector and the subjects on a scale from "None" to "Severe". Collection of adverse events and concomitant treatments during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins Dermscan, Villeurbanne, France